CLINICAL TRIAL: NCT05041998
Title: Improving Physical Function and Patient-reported Outcomes Through a Quantitatively-informed Socket Design Process
Brief Title: Quantitatively-informed Socket Design Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, William Anderst, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20070123; W81XWH2010914 (Other Grant/Funding Number: US Dept of Defense)
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Artificial Limbs

STUDY DESIGN:
Intervention Model Description: Participants will perform study activities with nine different versions (including the original unmodified) of their prosthetic socket in a randomized sequence.
Masking Description: The Research Technician and Engineer will be blinded to the socket modification when processing radiographic data from each trial. The participant will not be told the modification made to each socket, however the nature of the intervention (body worn prosthetic device) makes masking infeasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Unmodified Socket + 8 Socket Modifications in Random Order (Experimental): The sequence of the 9 different interventions (original socket and 8 versions derived from it) is randomized for each participant. The number of participants is smaller than the number of possible permutations. Therefore the enacted ordering is randomly selected from the pool of possible orderings. Participants walk for less than 10 minutes with every socket type while data is being collected.
  Interventions: Device: Trans-femoral prosthetic socket

INTERVENTIONS:
Device: Trans-femoral prosthetic socket — Unmodified) A custom-made check socket serving as the interface between residual limb and prosthesis
  1. Soft socket (Socket made from softer material than unmodified original)
  2. Stiff socket (Socket made from stiffer material than unmodified original)
  3. moderately lower brim height (Brim of the socket is lowered by 10% of socket length compared to unmodified original)
  4. slightly lower brim height (Brim of the socket is lowered by 5% of socket length compared to unmodified original)
  5. Oversized socket (The socket volume is 6% larger than the unmodified original)
  6. Undersized socket (The socket volume is 6% smaller than the unmodified original)
  7. CAT-CAM influenced geometry (The cross sectional geometry of the socket is modelled following the contoured adducted trochanteric-controlled alignment method (CAT-CAM))
  8. MAS influenced geometry (The cross sectional geometry of the socket is modelled following the Marlo Anatomic Socket (MAS) template)

SUMMARY:
This study will investigate the effects of specific standardized modifications to trans-femoral prosthetic sockets in a randomized within-subject design. This is in preparation for a subsequently planned clinical trial to validate the findings by implementing them into a fitting method for individual sockets.

DETAILED DESCRIPTION:
Background: Lower limb amputees experience chronic health challenges such as residual limb skin problems, low back pain, and osteoarthritis. These problems are exacerbated by high physical activity levels and by poor prosthetic socket fit. Prosthetists believe that limiting residual femur and skin motion will improve force coupling and thereby address these problems. However, there are no data demonstrating how changes in socket design affect residual femur and skin motion, and, by extension, lead to improved patient-reported outcomes.

Objective/Hypothesis: Goal of this research is to improve the current socket design optimization process that involves trial and error and relies heavily on the prosthetist's experience and intuition by using a quantitatively informed optimization process. The hypothesis is that modifiable in-socket mechanics, i.e. residual femur motion, skin strain, and pressure within the socket, are related to socket design and patient outcomes, and can be estimated using readily available clinical measurements.

Specific Aims: First aim is to identify the key characteristics of in-socket mechanics that are related to physical function and patient-reported comfort and function. The second aim is to identify readily available clinical measurements that are associated with the in-socket mechanical characteristics that are related to outcomes. The purpose of this aim is to correlate our laboratory findings from Aim 1 with more conventional modalities for clinical assessment.

Research Strategy: Preliminary data demonstrates the feasibility of the proposed research plan and will progress to a pilot clinical trial. The two aims will involve 30 transfemoral amputees. A highspeed biplane radiography system is used to image the residual limb while participants walk on a dual-belt instrumented treadmill both in their current socket and in sockets with purposely altered volume, brim height, cross-sectional geometry, and stiffness. Three-dimensional (3D) skin motion within the socket will be determined by tracking the motion of 40 to 50 small metal beads placed in a grid pattern on the skin of the residual limb before donning the socket. Residual femur motion within the socket will be determined with submillimeter accuracy using a validated tracking process that matches subject-specific bone models obtained from CT to the biplane radiographs. Discrete in-socket pressure will be recorded at four locations using pressure sensing pads. Readily available clinical measurements will be collected as well, including gait analysis, foot loading patterns, ground reaction forces, residual limb tissue stiffness, and hip range of motion hip strength. Each participant will complete clinical questionnaires to qualitatively evaluate comfort, fit, and overall satisfaction after wearing each socket. The different socket modifications are intended to affect the in-socket mechanics of the residual limb, physical function and patient-reported outcomes (Aim 1). These relationships will be assessed using a generalized linear model. Correlation between the research grade measurements and accessible clinical measures (Aim 2) will be evaluated using bivariate correlation analyses. The information gained in Aims 1 and 2 will be used to develop a quantitatively-informed socket optimization process, wherein the clinical measurements associated with in-socket mechanics will be used to inform socket design optimizations.

ELIGIBILITY:
Inclusion Criteria:

* Transfemoral prosthesis user
* 18-80 years of age
* Body weight less than 125 kg
* Able to walk unassisted on a treadmill

Exclusion Criteria:

* Pregnant females
* Clinically diagnosed osteoporosis
* Previous high exposure to radiation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Residual Femur motion | 1 second
  medial-lateral and superior-inferior translation of the distal femur relative to the socket from late swing through midstance
Skin strain | 1 second
  average and peak skin strain within each of four regions, expressed as a percentage of the gait cycle
Socket pressure | 20 seconds
  measure peak pressure and area under the pressure versus time curve, expressed as a percentage of the gait cycle

SECONDARY OUTCOMES:
Gait symmetry | 20 seconds
  average of the peak trunk lean, and the average peak hip flexion and extension, measured by motion capture system
Plantar pressure | 20 seconds
  peak plantar pressure from foot strike to midstance
Static displacement | 1 second
  distance from the most distal point of the residual femur to the inside surface of the socket under weightbearing
Tissue Stiffness | 3 seconds
  Average tissue stiffness for four regions of the residual limb
Trunk lean | 20 seconds
  Body angles based on markers placed on the shoulders and spine
Hip flexion/extension | 20 seconds
  Based on markers at greater trochanters, knee, ankle and foot.
Hip strength | 20 seconds
  Manual muscle testing of hip flexors and extensors
Hip Range of Motion | 20 seconds
  Manually measured using goniometer

CONTACTS AND LOCATIONS:
Overall Officials: William Anderst, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Delatorre Orthotics & Prosthetics, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other researchers at Pitt in the future
Supporting Information: Study Protocol, SAP, ICF
Time Frame: upon conclusion of the study (in 2025) with no expiration
Access Criteria: commensurate with applicable restrictions posed by the study sponsor

REFERENCES:
- [Derived] Anderst W, Fiedler G, Onishi K, McKernan G, Gale T, Paulus P. Within-subject effects of standardized prosthetic socket modifications on physical function and patient-reported outcomes. Trials. 2022 Apr 12;23(1):299. doi: 10.1186/s13063-022-06205-z. PMID 35413866